CLINICAL TRIAL: NCT04851444
Title: A Phase I Clinical Study on the Safety, Tolerability and Pharmacokinetics of SI-F019 Recombinant Human Bivalent ACE2-Fc Fusion Protein Injection in a Single Dose in Healthy Subjects
Brief Title: A Study of SI-F019 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI-F019-101
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SI-F019 (Experimental): SI-F019 administered intravenously (IV).
  Interventions: Drug: SI-F019

INTERVENTIONS:
Drug: SI-F019 — Single dose is administered IV.

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetic properties of a single intravenous administration of SI-F019 recombinant human bivalent ACE2-Fc fusion protein injection in healthy participants, and provide a basis for the design of subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. The participants fully understand the purpose, character, methods and possible adverse events of the trial, and volunteer to be the subject, and sign the informed consent form before the start of any study procedure, and guarantee that any procedure will be participated in the study by the participants themselves;
2. The participant could communicate well with the investigator, and understand and comply with the requirements of this study.
3. The participant has no history of chronic diseases or serious diseases such as cardiovascular, liver, kidney, breathing, blood and lymph, endocrine, immune, mental, nervous, gastrointestinal system, and is in good general health;
4. The participants (including male subjects) have no pregnancy plan and voluntarily take effective contraceptive measures during the screening period and within the next 6 months, and no sperm or egg donation plan, in which non-drug contraceptive measures should be used voluntarily during the trial period;
5. Male or female subjects aged 18 to 45 (including 18 and 45 years old);
6. Male weight ≥50.0 kg, female weight ≥45.0 kg; body mass index (BMI) is in the range of 19.0~26.0 kg/m2 (including cut-off value);
7. Vital signs examination, physical examination, clinical laboratory examination (blood routine, urine routine, blood biochemistry, blood transfusion, blood coagulation function, pregnancy test (female), alcohol and drug screening, etc.), 12-lead electrocardiogram and Abdominal B-ultrasound examination showed no abnormalities or abnormalities without clinical significance.

Exclusion Criteria:

1. Health condition: clinically significant medical history of heart, liver, kidney, digestive tract, nervous system, respiratory system, blood and lymph system, immune system, mental and metabolic abnormalities, and bones;
2. Those who have a history of allergies to biological agents or any drug component; those who have a history of allergies and are judged not to be included in the group by the investigator;
3. Those who have undergone surgery within 3 months before screening, or who plan to undergo surgery during the study period, and those who have undergone surgery that will affect drug absorption, distribution, metabolism, and excretion;
4. Those who cannot tolerate venipuncture or have a history of fainting needles and bleeding;
5. Those who have a history of drug abuse within 6 months before screening;
6. Used drugs within 3 months before screening;
7. Those who donated blood including blood components or a large amount of blood loss (≥200mL) within 3 months before screening, received blood transfusion or used blood products;
8. The participant (female) is in pregnancy or lactation during the screening period or the test process;
9. The participant has a birth plan or sperm donation or egg donation plan during the screening period and the next 6 months;
10. Those who have used any prescription drugs, over-the-counter drugs, and Chinese herbal medicines within 2 weeks before screening;
11. Those who have received vaccination within 4 weeks before screening, or plan to receive vaccination during the study period;
12. Those who smoked more than 5 cigarettes per day in the 3 months before screening, or who could not stop using any tobacco products during the trial period;
13. Drinking more than 14 units per week in the 3 months before screening (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine), or those who cannot abstain from alcohol during the test;
14. Those who have special requirements for diet and cannot accept a unified diet;
15. Those who have participated in drug clinical trials and used trial drugs within 3 months before screening;
16. Received immunosuppressive agents or monoclonal antibodies before screening;
17. For patients with abnormal vital signs that have clinical significance, refer to the normal range (including cut-off values): sitting systolic blood pressure 90~139mmHg, diastolic blood pressure 60~89mmHg, pulse 60-100 beats/min, body temperature (ear temperature) 35.4~37.7℃, breathing 16-20 times/min, the specific situation will be judged comprehensively by the investigator;
18. Any abnormality in laboratory examinations and auxiliary examinations, and the investigator judges that it has clinical significance;
19. One or more of hepatitis B virological indicators, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody test has one or more clinical significance;
20. Female participants who have a positive urine or blood pregnancy test result during the screening period;
21. Alcohol breath test results greater than 0.0mg/100mL or drug screening positive (morphine, methamphetamine, ketamine, ecstasy (dimethyldioxyamphetamine), cannabis (tetrahydrocannabinolic acid);
22. Acute illness occurred during the period from screening to -1 day of admission;
23. Those who have taken any prescription drugs, over-the-counter drugs, or Chinese herbal medicines during the period from screening to -1 day of admission;
24. The investigator determines that the participant is not suitable for the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
SAE | Up to 29 days after the first dose of SI-F019
  Number of Adverse Events and Seriuos Adverse Events

SECONDARY OUTCOMES:
Tmax | 7 days
  Maximum Time
t1/2 | 7 days
  half time

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Principal Investigator — Shanghai Public Health Clinical Center Ethics Committee Approval Letter
Locations (1):
- Shanghai Public Health Clinical Center Ethics Committee Approval Letter, Shanghai, Shanghai Municipality, China